CLINICAL TRIAL: NCT00621881
Title: A Phase 1, Repeated-Dose, Open-Label Study to Investigate the Pharmacokinetics and Safety of Naproxcinod 750 mg Bid Administered to Patients With Impaired Hepatic Function Compared to Matching Healthy Subjects
Brief Title: A Phase 1 Study to Compare the PK and Safety of Naproxcinod in Hepatic Impaired Patients and Matching Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NicOx (Industry)
Responsible Party: Dr Brigitte Duquesroix, Senior Director of Clinical Research, nicox
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HCT3012-X-105
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2011-06

CONDITIONS: Liver Disease
Keywords: hepatic impairment
MeSH Terms: conditions — Liver Diseases | interventions — naproxen-n-butyl nitrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): 750 mg naproxcinod
  Interventions: Drug: naproxcinod

INTERVENTIONS:
Drug: naproxcinod — 750 mg bid

SUMMARY:
This is an open-label study that will compare the pharmacokinetic and safety effects of naproxcinod in hepatic impaired patients vs. matching healthy subjects.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, parallel-group study that will be conducted at two study sites. Patients with hepatic impairment and matched healthy subjects will receive naproxcinod 750 mg bid for 6 days and qd for the last day.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, age 40 to 75 years with stable hepatic insufficiency conforming to Child-Pugh classification B OR
* Male or Female, age 40 to 75 years with similar distribution of age, weight, gender, smoking habits, and race, and in general good health

Exclusion Criteria:

* Current or expected use of anticoagulants or analgesic, anti-inflammatory therapies except lose dose aspirin
* History of renal impairment
* Diagnosis of gastric or duodenal ulceration and/or history of significant gastro-duodenal bleeding within the last 6 months
* Clinically relevant abnormal ECG
* Alcohol or drug abuse within the last 6 months
* Any significant or chronic disease (except hepatic insufficiency for the patient cohort) which may interfere with study evaluations

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
To assess the pharmacokinetics of naproxcinod and its metabolites after repeated 750 mg bid oral administration of naproxcinod in hepatic impaired patient in comparison with matching healthy subjects | 8 days

SECONDARY OUTCOMES:
To assess safety and tolerability of repeated 750 mg bid oral administration of naproxcinod in hepatic impaired patients in comparison with matching healthy subjects. | 8 days

CONTACTS AND LOCATIONS:
Locations (1):
- Miami, Florida, United States